CLINICAL TRIAL: NCT03885089
Title: Infliximab BS for Intravenous Drip Infusion 100 mg "Pfizer" General Investigation (Psoriasis Vulgaris, Psoriasis Arthropathica, Pustular Psoriasis, or Erythrodermic Psoriasis)
Brief Title: Infliximab Biosimilar for Intravenous Drip Infusion 100 mg "Pfizer" Drug Use Investigation (Psoriasis)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B5371009; NCT03885089 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2019-03-04; First posted 2019-03-21 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis Vulgaris; Psoriasis Arthropathica; Pustular Psoriasis; Erythrodermic Psoriasis
Keywords: Infliximab; biosimilar
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab [infliximab biosimilar 3]: Patients with Psoriasis Vulgaris, Psoriasis Arthropathica, Pustular Psoriasis, or Erythrodermic Psoriasis treated by Infliximab BS
  Interventions: Drug: Infliximab [infliximab biosimilar 3]

INTERVENTIONS:
Drug: Infliximab [infliximab biosimilar 3] — <Psoriasis> The usual dose is 5 mg as Infliximab (Genetical Recombination) [Infliximab Biosimilar 3] for every kg of body weight given as an intravenous infusion. After an initial dose is given, the subsequent doses are given at Weeks 2 and 6, and every 8 weeks thereafter. After a dose at Week 6 is given, the dose may be increased or the dosing interval may be reduced for patients who have an incomplete response or reduced effects. These adjustments should be made in a stepwise manner according to condition of patients. The maximum dose is 10 mg for every kg of body weight at the dosing interval of 8 weeks and 6 mg for every kg of body weight at a reduced dosing interval. The minimum dosing interval is 4 weeks.
  Other Names: Infliximab BS for Intravenous Drip Infusion 100 mg "Pfizer"

SUMMARY:
To collect information on the safety and effectiveness of Infliximab BS for Intravenous Drip Infusion 100 mg "Pfizer" against psoriasis vulgaris, psoriasis arthropathica, pustular psoriasis, or erythrodermic psoriasis under actual status of use.

DETAILED DESCRIPTION:
This study will be conducted with all-case investigation system in patients with psoriasis vulgaris, psoriasis arthropathica, pustular psoriasis, or erythrodermic psoriasis.

This study will be conducted in patients who used this drug after the day of approval of dosage and administration for psoriasis at contracted medical institutions. Patients who used this drug before conclusion of the contract with the medical institution will also be included in this study (retrospective patients will be included).

Therefore, Time Perspective is retrospective and prospective.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis vulgaris, psoriasis arthropathica, pustular psoriasis, or erythrodermic psoriasis who started treatment with this drug
* Patients who received this drug for the first time at the medical institution after the day of launch of this drug.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Psoriasis Vulgaris, Psoriasis Arthropathica, Pustular Psoriasis, or Erythrodermic Psoriasis treated by Infliximab BS
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local Country Office, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5371009

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]: Participants with psoriasis vulgaris, psoriasis arthropathica, pustular psoriasis, or erythrodermic psoriasis who received Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] as indicated in the approved local product document for the first time were observed for 30 weeks from the day of initial dose of this drug. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Started | 10
Completed | 8
Not Completed | 2
Not completed — No informed consent for publication of study results | 2

BASELINE CHARACTERISTICS:
Population: A total of 10 participants were enrolled in this study. Of the 10 participants from whom case report forms were collected, 2 participants were excluded from the safety analysis set due to no informed consent for publication of study results.
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 8
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 5
  ≥65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was a treatment-related adverse event, and any untoward medical occurrence attributed to Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] in a participant who received this drug. A serious ADR was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Relatedness to Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] was assessed by the physician.
Time Frame: 30 weeks from the day of initial dose
Population: The safety analysis set (8 participants) comprised of participants who satisfied the inclusion criteria and had received Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]. Participants with no informed consent for publication of study results were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 8
Participants | 2

2. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI75) Response
Description: Percentage of participants with a PASI75 response was presented along with the two-sided 95% confidence interval (exact method).
  The PASI quantifies the severity of lesions and the percentage of lesion area. It is the total score of the degree of erythema, infiltration/thickening, and scaling (evaluated for each skin finding) in each of the 4 body regions evaluated by the physician. The score was adjusted for the percentage of lesion area of skin rash in each body region and the percentage of the area of each body region to the whole body. The percent change (%) in PASI score from baseline to the study completion date was calculated for each participant, and the number and proportion of participants with ≥ 75% improvement were calculated as PASI75.
Time Frame: 30 weeks from the day of initial dose
Population: The efficacy analysis set (4 participants) comprised of participants in the safety analysis set who had effectiveness evaluation. Of the 4 participants, percentage of participants with a PASI75 response as of the study completion date was calculated for the 3 participants whose PASI scores both at baseline and study completion date were available.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 3
Percentage of Participants | 0.0 [0.00 to 70.76]

3. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 90 (PASI90) Response
Description: Percentage of participants with a PASI90 response was presented along with the two-sided 95% confidence interval (exact method).
  The PASI quantifies the severity of lesions and the percentage of lesion area. It is the total score of the degree of erythema, infiltration/thickening, and scaling (evaluated for each skin finding) in each of the 4 body regions evaluated by the physician. The score was adjusted for the percentage of lesion area of skin rash in each body region and the percentage of the area of each body region to the whole body. The percent change (%) in PASI score from baseline to the study completion date was calculated for each participant, and the number and proportion of participants with ≥ 90% improvement were calculated as PASI90.
Time Frame: 30 weeks from the day of initial dose
Population: The efficacy analysis set (4 participants) comprised of participants in the safety analysis set who had effectiveness evaluation. Of the 4 participants, percentage of participants with a PASI90 response as of the study completion date was calculated for the 3 participants whose PASI scores both at baseline and study completion date were available.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 3
Percentage of Participants | 0.0 [0.00 to 70.76]

4. Secondary Outcome: Change From Baseline in Body Surface Area Involvement (BSA)
Description: Summary statistics of the BSA at baseline, at study completion date, and the change in BSA from baseline to study completion date was presented.
  BSA was calculated from the percentage of skin rash to body surface area from baseline to study completion date, and change in severity of disease was evaluated.
Time Frame: 30 weeks from the day of initial dose
Population: The efficacy analysis set (4 participants) comprised of participants in the safety analysis set who had effectiveness evaluation. Of the 4 participants, summary statistics and change from baseline in BSA as of the study completion date was calculated for the 1 participant whose BSA both at baseline and study completion date were available.
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 1
Percentage of BSA
  At baseline | 0.00 (NA) — The standard deviation was not available due to the small number of participants whose BSA was calculated.
  At study completion date | 30.00 (NA) — The standard deviation was not available due to the small number of participants whose BSA was calculated.
  Change | 30.00 (NA) — The standard deviation was not available due to the small number of participants whose BSA was calculated.

ADVERSE EVENTS:
Time Frame: 30 weeks from the day of initial dose
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both events during the study.
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] (N=8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT03885089/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT03885089/SAP_001.pdf